CLINICAL TRIAL: NCT03979612
Title: Evaluation of the Adhesion to the Network of Care of People at Genetic Risk of Cancer in Midi-Pyrénées (GENEPY)
Brief Title: Evaluation of the Adhesion to the GENEPY Network
Acronym: GENEPY
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Other Study IDs: 18HLGENE03
Record Dates: First submitted 2019-06-04; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Hereditary Cancer Syndrome; Hereditary Breast and Ovarian Cancer; Hereditary Colorectal Endometrial Cancer Syndrome
Keywords: breast; hereditary; cancer; ovarian; predisposition
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary; Hereditary Breast and Ovarian Cancer Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis; Neoplasms; Disease Susceptibility

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: inclusion of subjects in the GENEPY network — The inclusion of subjects in the GENEPY network follows the genealogical study of a case (index): relatives are identified as potentially at risk. In accordance with the recommendations, but also generally at the wish of the patients (Claes 2003), the index case is then asked to inform its relatives and to propose them to go to an oncogenetic consultation of their choice. If these people reside in the Midi Pyrenees Toulouse oncogenetic consultation is open to them. If following this consultation a mutation is identified or that their genetic risk is considered important, they are proposed to join the GENEPY network for their monitoring.

SUMMARY:
In order to best meet the needs of all those affected by the genetic risk of cancer in our region, it is important to identify the factors likely to influence the course leading to the GENEPY surveillance network. The aim of this study is to evaluatie the adhesion to the network of care of people at genetic risk of cancer in Midi-Pyrénées (GENEPY).

DETAILED DESCRIPTION:
This network has been open since November 2015 for people who are genetically predisposed to breast / ovarian cancer. The extension to digestive pathologies (HNPCC syndrome, PAF) is in progress. It concerns not only the persons carrying a mutation also those belonging to a family without identified mutation but whose risk of predisposition is important.

The GENEPY network is based on a collaboration between oncogenetic consultations in the region and professionals practicing in institutions (private, public) and liberal: general practitioners, gynecologists, radiologists, oncologists, gastroenterologists, psychologists ...

It is therefore a multicentric and multidisciplinary network, which aims to promote the local care of people genetically predisposed (or considered at high risk of genetic predisposition), while ensuring a high level of competence, to guarantee an optimal and equitable care on the whole of Midi Pyrenees.

The diagnosis of a new genetic disease in an individual is likely to have implications for other family members who may themselves be at risk of developing the disease and / or passing it on to their children.

The inclusion of subjects in the GENEPY network follows the genealogical study of a case (index) : relatives are identified as potentially at risk. In accordance with the recommendations, but also generally at the wish of the patients, the index case is then asked to inform its relatives and to propose them to go to an oncogenetic consultation of their choice. If these people reside in the Midi Pyrenees Toulouse oncogenetic consultation is open to them. If following this consultation a mutation is identified or that their genetic risk is considered important, they are proposed to join the GENEPY network for their monitoring.

ELIGIBILITY:
Inclusion Criteria:

* people with an identified mutation, predisposing to tumors of the breast / ovary or colon / rectum
* people resident in the Midi-Pyrénées region

Exclusion Criteria:

* people under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The inclusion of subjects in the GENEPY network follows the genealogical study of a case (index): relatives are identified as potentially at risk. In accordance with the recommendations, but also generally at the wish of the patients (Claes 2003), the index case is then asked to inform its relatives and to propose them to go to an oncogenetic consultation of their choice. If these people reside in the Midi Pyrenees Toulouse oncogenetic consultation is open to them. If following this consultation a mutation is identified or that their genetic risk is considered important, they are proposed to join the GENEPY network for their monitoring.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Adhesion to the GENEPY network | 6 months
  Network membership rate : comparison between the number of relatives who received the invitation and the number of them who joined the network.
Age of relatives | 1 day
  Age of the relative of the patient who answered the questionnaire
Sex of relatives | 1 day
  sex of the relative of the patient who answered the questionnaire
Place of residence of the relatives | 1 day
  distance from the offer of care and level of deprivation (for the relative of the patient who answered the questionnaire)
Proximity to the index case | 1 day
  relationship of the relatives with the index case according to the latter contact
Cancer status Communication | 1 day
  Patient's agreement to communicate about his illness to his relative

SECONDARY OUTCOMES:
People satisfaction | 1 year
  satisfaction of people who have joined the network (scale of values by questionnaire)
Practionners satisfaction | 1 year
  satisfaction of general practitioners (scale of values by questionnaire)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Claudius Regaud - IUCT-Oncopole, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eisinger F, Bressac B, Castaigne D, Cottu PH, Lansac J, Lefranc JP, Lesur A, Nogues C, Pierret J, Puy-Pernias S, Sobol H, Tardivon A, Tristant H, Villet R. [Identification and management of hereditary breast-ovarian cancers (2004 update)]. Pathol Biol (Paris). 2006 May;54(4):230-50. doi: 10.1016/j.patbio.2006.02.002. Epub 2006 May 2. French. PMID 16632260
- [Result] Landsbergen K, Verhaak C, Kraaimaat F, Hoogerbrugge N. Genetic uptake in BRCA-mutation families is related to emotional and behavioral communication characteristics of index patients. Fam Cancer. 2005;4(2):115-9. doi: 10.1007/s10689-004-7991-2. PMID 15951961
- See also: General information from National Institue for Cancer (INCa) — http://www.e-cancer.fr/Professionnels-de-sante/Recommandations-et-outils-d-aide-a-la-pratique/Oncogenetique-ou-Cancers-avec-predispositions-genetiques
- Available data/document: Individual Participant Data Set — https://www.iuct-oncopole.fr/information-sur-les-donnees-de-sante — General information on our web site about investigations from patients data